CLINICAL TRIAL: NCT01500356
Title: Effect of Exercise and Weight Loss on Cardiovascular Health
Acronym: Heart Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, John M. Jakicic, PhD, PhD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HL103646
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Cardiovascular Disease; Obesity
Keywords: cardiovascular disease; obesity; exercise
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Motor Activity | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Diet alone (Experimental): Weight loss intervention that focuses only on reducing energy intake of the diet.
  Interventions: Behavioral: Behavioral weight loss intervention
- Diet plus Moderate Exercise (Experimental): Weight loss intervention that involve an energy restricted diet (identical to the Diet Alone arm) plus the inclusion of 150 minutes per week of moderate-intensity exercise.
  Interventions: Behavioral: Diet Plus Moderate Exercise
- Diet Plus High Exercise (Experimental): Weight loss intervention that involve an energy restricted diet (identical to the Diet Alone arm) plus the inclusion of 250-300 minutes per week of moderate-intensity exercise.
  Interventions: Behavioral: Diet Plus High Exercise

INTERVENTIONS:
Behavioral: Behavioral weight loss intervention — Weight loss intervention that focuses on reducing energy intake.
  Arms: Diet alone
Behavioral: Diet Plus Moderate Exercise — Weight loss intervention that involve an energy restricted diet (identical to the Diet Alone arm) plus the inclusion of 150 minutes per week of moderate-intensity exercise.
  Arms: Diet plus Moderate Exercise
Behavioral: Diet Plus High Exercise — Weight loss intervention that involve an energy restricted diet (identical to the Diet Alone arm) plus the inclusion of 250-300 minutes per week of moderate-intensity exercise.
  Arms: Diet Plus High Exercise

SUMMARY:
The primary aim of this study is to examine the effect of the consensus public health recommended level of physical activity [moderate physical activity (MOD-PA) = 150 min/wk] versus a higher dose of physical activity [high physical activity (HIGH-PA) = 250 min/wk] in the context of a comprehensive behavioral weight loss program that a includes a reduction in energy intake measures of cardiovascular function using cardiac MRI and biomarkers of vascular disease risk. Each of these exercise doses will be compared independently to a Diet Only group intervention on the proposed primary and secondary outcomes, with MOD-PA also compared to HIGH-PA. This study involves the recruitment of 390 overweight and obese adults who will be randomly assigned to one of the above conditions (Diet Only, MOD-PA, HIGH-PA) for a period of 12 months. The primary outcome is LVM measured by cardiac MRI. Secondary outcomes include additional cardiac MRI measures (aortic pulse wave velocity, end diastolic volume, aortic distensibility), inflammatory markers (CRP and TNFα) and selected adipocytokines (adiponectin) as biomarkers of risk related to vascular outcomes, body weight, body composition, and cardiorespiratory fitness, and traditional CVD risk factors (lipids, glucose, insulin, blood pressure). Additional secondary analyses will allow for examination of the effects of physical activity independent of weight change on the primary and secondary outcomes.

DETAILED DESCRIPTION:
Current estimates indicate that in excess of 65 percent of adults in the United States are overweight (BMI >25.0 kg/m2) with at least 30 percent of adults classified as obese (BMI >30 kg/m2). Overweight and obesity have been linked to numerous chronic conditions including cardiovascular disease. The application of cardiac MRI (CMRI) allows for direct measurement of the cardiac structure, and left ventricular mass (LVM) assessed by CMRI has been shown to be predictive of cardiovascular disease. Recent studies have shown that LVM is decreased with weight loss; however, there is a lack of information on the added benefit of physical activity to weight loss on these direct measures of cardiovascular structure and function. Thus, consistent with PA-09-243, this study will examine the effect of two recommended doses of physical activity combined with a dietary intervention on changes in the proposed outcomes of cardiovascular disease risk in overweight adults.

The primary aim of this study is to examine the effect of the consensus public health recommended level of physical activity [moderate physical activity (MOD-PA) = 150 min/wk] versus a higher dose of physical activity [high physical activity (HIGH-PA) = 250 min/wk] in the context of a comprehensive behavioral weight loss program that a includes a reduction in energy intake measures of cardiovascular function using cardiac MRI and biomarkers of vascular disease risk. Each of these exercise doses will be compared independently to a Diet Only group intervention on the proposed primary and secondary outcomes, with MOD-PA also compared to HIGH-PA. This study involves the recruitment of 390 overweight and obese adults who will be randomly assigned to one of the above conditions (Diet Only, MOD-PA, HIGH-PA) for a period of 12 months. The primary outcome is LVM measured by cardiac MRI. Secondary outcomes include additional cardiac MRI measures (aortic pulse wave velocity, end diastolic volume, aortic distensibility), inflammatory markers (CRP and TNFα) and selected adipocytokines (adiponectin) as biomarkers of risk related to vascular outcomes, body weight, body composition, and cardiorespiratory fitness, and traditional CVD risk factors (lipids, glucose, insulin, blood pressure). Additional secondary analyses will allow for examination of the effects of physical activity independent of weight change on the primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age.
* Body mass index (BMI) between 25.0 to <40.0 kg/m2.
* Ability to provide informed consent prior to participation in this study.

Exclusion Criteria:

* Females who are currently pregnant or breastfeeding, or reporting that she is planning a pregnancy within the next 12 months.
* History of bariatric surgery.
* Report current medical condition or treatment for a medical condition that could affect body weight. These may include the following: cancer (Note: Persons previously diagnosed with non-melanoma skin cancers, those successfully treated for cancer who have remained disease-free for five years or more would be eligible for participation in this study); diabetes mellitus; hyperthyroidism; inadequately controlled hypothyroidism; chronic renal insufficiency; chronic liver disease; gastrointestinal disorders including ulcerative colitis, Crohn's disease, or malabsorption syndromes; etc.
* Current congestive heart failure, angina, uncontrolled arrhythmia, symptoms indicative of an increased acute risk for a cardiovascular event, prior myocardial infarction, coronary artery bypass grafting or angioplasty, conditions requiring chronic anticoagulation (i.e. recent or recurrent DVT).
* Resting systolic blood pressure of >160 mmHg or resting diastolic blood pressure of >100 mmHg.
* Eating disorders that would contraindicate weight loss or physical activity.
* Alcohol or substance abuse.
* Currently treated for psychological issues (i.e., depression, bipolar disorder, etc), taking psychotropic medications within the previous 12 months, or hospitalized for depression within the previous 5 years.
* Report exercise on >3 days per week for >20 minutes per day over the past 3 months. (NOTE: It is important that individuals are sedentary when entering this study to allow for maximal effect of the intervention.)
* Report weight loss of >5% or participating in a weight reduction diet in the past 3 months.
* Report plans to relocate to a location not accessible to the study site or having employment, personal, or travel commitments that prohibit attendance to at least 80 percent of the scheduled intervention sessions and all of the scheduled assessments.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 383 (Actual)
Dates: Start 2011-12-13 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Left ventricular mass assessed using cardiac MRI | Baseline (0 months) and 12 months
  Left ventricular mass will be assessed using cardiac MRI

SECONDARY OUTCOMES:
Change in end-diastolic volume assessed using cardiac MRI | baseline (0 months) and 12 months
  Assessed using cardiac MRI
Change in cardiorespiratory fitness | baseline (0 months) 6 months, and 12 months
  Measured using a graded exercise test
Change in blood levels of C-Reactive Protein (CRP) | baseline (0 months), 6 months, and 12 months
  Assessed from a fasting blood sample
Change in body weight | baseline (0 months), 6 months, and 12 months
Change in body composition | baseline (0 months), 6 months, and 12 months
  Measured using dual-energy x-ray absorptiometry (DXA)
Change in regional adiposity | baseline (0 months), 6 months, 12 months
  Measured using anthromometry that includes girth measures of the waist and hip
Change in physical activity | baseline (0 months), 6 months, 12 months
  Measured using both a wearable device and by questionnaire
Change in energy intake | baseline (0 months), 6 months, 12 months
  Assessed using a questionnaire
Change in traditional CVD risk factors (lipids, glucose, insulin) | baseline (0 months), 6 months, 12 months
  Measured from a fasting blood sample
Change in resting blood pressure | baseline (0 months), 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: John M. Jakicic, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Jakicic JM, Rogers RJ, Lang W, Gibbs BB, Yuan N, Fridman Y, Schelbert EB. Impact of weight loss with diet or diet plus physical activity on cardiac magnetic resonance imaging and cardiovascular disease risk factors: Heart Health Study randomized trial. Obesity (Silver Spring). 2022 May;30(5):1039-1056. doi: 10.1002/oby.23412. PMID 35470972